CLINICAL TRIAL: NCT06359145
Title: Prediction of COPD Chest CT Severity Using Electrical Impedance Tomography by Machine Learning Methods
Brief Title: Prediction of COPD Severity Using Electrical Impedance Tomography
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Director, Department of Respiratory and Critical Care Medicine, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: EIT and COPD
Record Dates: First submitted 2024-03-30; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Electric Impedance; Respiratory Function Tests; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to predict the CT visual score of emphysema with EIT-based parameters, in order to provide a non-invasive and convenient method for the evaluation of lung structure and physiological and pathological progression of COPD.

DETAILED DESCRIPTION:
Methods: By collecting pulmonary function data, CT visual scores, and EIT data, and employing deep machine learning algorithms to compare the predictive capabilities of EIT and PFT for CT visual scores of pulmonary emphysema, this study aims to validate the ability of EIT to assess the progression of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical physicians suspect a patient may have COPD based on symptoms and physical examination, but a definitive diagnosis has not been confirmed through PFTs.
* Age > 20 years, and be able to communicate with doctors.
* Willing to sign informed consent for the course of the study.

Exclusion Criteria:

* Patient refusal of EIT examination.
* The CT scan information is incomplete, and the interval between the pulmonary function test and the CT scan is more than 180 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical physicians suspect a patient may have COPD based on symptoms and physical examination, but a definitive diagnosis has not been confirmed through PFTs.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The predictive power of EIT and PFT for CT visual scoring of emphysema | 1 mounths
  the prediction accuracy between deep machine learning models based on PFT data and EIT data

CONTACTS AND LOCATIONS:
Locations (1):
- PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No